CLINICAL TRIAL: NCT01404234
Title: Open-Label Phase 3 Trial to Evaluate the Safety of Aztreonam 75 mg Powder and Solvent for Nebuliser Solution/Aztreonam for Inhalation Solution (AZLI) in Children With Cystic Fibrosis (CF) and Chronic Pseudomonas Aeruginosa (PA) in the Lower Airways
Brief Title: Safety of AZLI in Children With Cystic Fibrosis (CF) and Chronic Pseudomonas Aeruginosa in the Lower Airways
Acronym: PALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-205-0160
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa
Keywords: Cystic fibrosis; CF; PA; Pseudomonas aeruginosa; AZLI; aztreonam; Chronic Pseudomonas aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Aztreonam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label AZLI (Experimental): Participants received three 28-day courses of AZLI, each followed by 28 days off-treatment.
  Interventions: Drug: AZLI

INTERVENTIONS:
Drug: AZLI — AZLI 75 mg was administered 3 times daily via the investigational nebulizer.
  Other Names: Cayston®

SUMMARY:
This was an open-label, multicenter study in children ≤ 12 years of age with cystic fibrosis (CF) and chronic Pseudomonas aeruginosa (PA) infection in the lower airways using three 28-day courses of Aztreonam for Inhalation Solution (AZLI) 75 mg three times daily, each followed by 28 days off AZLI. The total treatment duration was to be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as determined by the 1997 CF Consensus Conference criteria:

  * Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test OR
  * Abnormal nasal transepithelial potential difference (NPD) test OR
  * A genotype with 2 identifiable mutations consistent with CF AND
  * One or more clinical features consistent with CF.
* Documented positive lower respiratory tract culture for PA at the screening visit plus two documented positive lower respiratory tract cultures for PA within 12 months prior to study entry (must have been a minimum 3 months apart.)
* Clinically stable with no evidence of significant respiratory symptoms or, if obtained for clinical evaluation, no chest radiograph findings at screening that would have required administration of IV antipseudomonal antibiotics, oxygen supplementation, or hospitalization.

Exclusion Criteria:

* Use of IV or inhaled antipseudomonal antibiotics within 14 days of study entry
* Presence of a condition or abnormality that would have compromised the participant's safety or the quality of study data, in the opinion of the investigator
* History of sputum or throat swab culture yielding Burkholderia spp. within 2 years prior to screening visit
* History of hypersensitivity/adverse reaction to aztreonam
* History of hypersensitivity/adverse reaction to beta-agonists
* History of lung transplantation
* Administration of any investigational drug or device within 30 days prior to screening visit or within 6 half-lives of the investigational drug (whichever was longer)
* Hospitalization for pulmonary-related illness within 28 days prior to screening visit
* Changes in or initiation of chronic azithromycin treatment within 28 days prior to screening visit
* Changes in or initiation of hypertonic saline treatment within 7 days prior to screening visit; for subjects on a stable regimen of hypertonic saline (28 days on/28 days off), beginning or ending a cycle of hypertonic saline was allowed
* Changes in antimicrobial, bronchodilator (BD), corticosteroid or dornase alfa medications within 7 days prior to screening visit;
* Changes in physiotherapy technique or schedule within 7 days prior to screening visit
* Abnormal renal or hepatic function results at most recent test within the previous 90 days

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bresnik, M.D., Study Director — Gilead Sciences
Locations (29):
- United States (10):
  - The Children's Hospital - Denver, Aurora, Colorado
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Mercy Hospital & Clinics, Kansas City, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- France (3):
  - C.H.U de Bordeaux, Bordeaux
  - Centre Hospitalier Robert Bissons, Lisieux
  - Hopital Necker Enfants Malades, Paris
- Germany (5):
  - Charite Campus Virchow Klinikum, Berlin
  - Universitatsklinik St. Josef-Hospital, Bochum
  - Kinder und Jugendklinik, Abteilung Lungen Bronchialheikunde, Erlandgen
  - Universitatsklinikum Essen, Essen
  - J.W. Goethe University Hopsital, Frankfurt
- Italy (3):
  - Azienda Ospedaliero Universitaria - Policlinico di Catania, Catania
  - A. Meyer Children Hospital Florence, Florence
  - Azienda Ospedaliera Instituti Ospitalieri di Verona, Verona
- Poland (3):
  - Specjalistyczny Zespot Opieki Zdrowotnej nad Matka i Dzieckiem, Gdansk
  - Instytut Gruzlicy I Chorob Pluc, Rabka-Zdrój
  - Instytut Matki i Dziecka, Warsaw
- Spain (5):
  - Pediatric Pneunmonology and Cystic Fibrosis Clinic, Barcelona
  - Hospital Infantil La Paz, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hosp. Mat-Inf. Carlos Haya, Málaga

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a total of 25 study sites in the United States and Europe. The first participant was screened on 29 December 2011. The last participant observation was on 03 April 2013.
Pre-assignment Details: 74 participants were screened; 61 participants were enrolled and treated, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- AZLI: Participants received three 28-day courses of Aztreonam for Inhalation Solution (AZLI), each followed by 28 days off-treatment. AZLI 75 mg was administered 3 times daily via the investigational nebulizer.
Period: Overall Study
Arm/Group | AZLI
Started | 61
Completed | 59
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- AZLI: Participants received three 28-day courses of AZLI, each followed by 28 days off-treatment. AZLI 75 mg was administered 3 times daily via the investigational nebulizer.
Arm/Group | AZLI
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (2.94)
Age, Customized [Number; unit: participants]
  < 2 years | 2
  ≥ 2 years to < 6 years | 7
  ≥ 6 years to ≤ 12 years | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African Heritage | 2
  White | 55
  Other | 3
  Not Permitted | 1
Region of Enrollment [Number; unit: participants]
  France | 5
  United States | 29
  Spain | 5
  Poland | 11
  Germany | 5
  Italy | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 16.3 (1.66)
Forced expiratory volume in 1 second (FEV1) % predicted [Mean (Standard Deviation); unit: percentage of FEV1 % predicted] — FEV1 % predicted is defined as FEV1 of the patient divided by the average FEV1 in the population for any person of similar age, sex, race, and body composition. Participants ≥ 6 years of age were analyzed at baseline for FEV1 % predicted (n = 52).
  percentage of FEV1 % predicted | 80.31 (19.494)
FEV1 [Mean (Standard Deviation); unit: liters] — FEV1 is defined as the maximal volume of air that can be exhaled in 1 second. Participants ≥ 6 years of age were analyzed at baseline for FEV1 (n = 52).
  liters | 1.67 (0.627)
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: liters] — FVC is defined as the volume of air that can forcibly be blown out after taking a full breath. Participants ≥ 6 years of age were analyzed at baseline for FVC (n = 52).
  liters | 2.11 (0.687)
FEV25-75 [Mean (Standard Deviation); unit: liters/sec] — FEF25-75 is defined as the forced expiratory flow from 25% to 75% of the FVC. Participants ≥ 6 years of age were analyzed at baseline for FEV25-75 (n = 52).
  liters/sec | 1.82 (1.169)
CFQ-R RSS Score [Mean (Standard Deviation); unit: units on a scale] — Respiratory symptoms (eg, coughing, congestion, wheezing) were assessed with the Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS). The range of scores (units) was 0 to 100 with higher scores indicating fewer symptoms. Participants ≥ 6 years of age were analyzed at baseline for CFQ-R RSS (n = 51; data was missing for one participant).
  units on a scale | 71.73 (17.327)
Presence of Pseudomonas aeruginosa (PA) [Number; unit: participants]
  Present | 58
  Absent | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to Safety or Tolerability Reasons
Description: Participants who discontinued study drug due to safety or tolerability reasons were defined as those with "Adverse Event (AE)/Safety or Tolerability" on the Study Drug Completion electronic case report form as the reason for early discontinuation. The 95% confidence interval (CI) was calculated using the exact binomial method.
Time Frame: Baseline to Day 168
Population: Participants in the Full Analysis Set (enrolled and received at least 1 dose of study medication) who completed the study or discontinued study drug due to safety or tolerability reasons were analyzed. Two participants voluntarily withdrew from the study prior to completion (not due to AEs/safety or tolerability reasons).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 59
percentage of participants | 0.0 [0.0 to 6.1]

2. Secondary Outcome: Change From Baseline in FEV1 % Predicted in Subjects Aged ≥ 6 Years
Description: The change in FEV1 % predicted was assessed at the end of each 28-day AZLI treatment course.
  FEV1 % predicted is defined as FEV1 of the patient divided by the average FEV1 in the population for any person of similar age, sex, race, and body composition.
Time Frame: Baseline to Day 28, 84, and 140
Population: Participants in the Full Analysis Set ≥ 6 years of age were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of FEV1 % predicted
Arm/Group | AZLI
Number analyzed (Participants) | 52
percentage of FEV1 % predicted
  Change at Day 28 (on-treatment, n = 52) | 4.73 (11.703)
  Change at Day 84 (on-treatment, n = 51) | 1.72 (12.516)
  Change at Day 140 (on-treatment, n = 50) | 1.65 (10.340)

3. Secondary Outcome: Change From Baseline in CFQ-R Respiratory Symptoms Scale (RSS) Score in Subjects Aged ≥ 6 Years
Description: The change in CFQ-R RSS score was assessed at the end of each 28-day AZLI treatment course.
  The range of scores (units) was 0 to 100 with higher scores indicating fewer symptoms.
Time Frame: Baseline to Day 28, 84, and 140
Population: Participants in the Full Analysis Set ≥ 6 years of age were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI
Number analyzed (Participants) | 52
units on a scale
  Change at Day 28 (on-treatment, n = 51) | 8.66 (14.903)
  Change at Day 84 (on-treatment, n = 48) | 9.38 (18.243)
  Change at Day 140 (on-treatment, n = 48) | 5.90 (15.372)

4. Secondary Outcome: Change in Pseudomonas Aeruginosa (PA) Sputum Density
Description: The change in PA sputum density (log10 colony-forming units per gram [cfu/g]) was assessed at the end of each 28-day AZLI treatment course.
Time Frame: Baseline to Day 28, 84, and 140
Population: Participants in the Full Analysis Set ≥ 6 years of age were analyzed.
Measure: Mean (Standard Deviation); unit: log10 CFU/g
Arm/Group | AZLI
Number analyzed (Participants) | 61
log10 CFU/g
  Change at Day 28 (on-treatment, n = 24) | -2.6 (2.50)
  Change at Day 84 (on-treatment, n = 25) | -2.0 (2.14)
  Change at Day 140 (on-treatment, n = 23) | -1.2 (2.13)

5. Secondary Outcome: Percentage of Participants Who Used Additional (Non-study) Antipseudomonal Antibiotics
Description: The percentage of participants who used additional (non-study) antipseudomonal antibiotics (IV, inhaled, oral, IV/inhaled, IV/inhaled/oral) was summarized (number and percent) for all subjects.
Time Frame: Baseline to Day 168
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 61
percentage of participants
  Never used non-study antipseudomonal antibiotics | 42.6
  Used non-study antipseudomonal antibiotics | 57.4

6. Secondary Outcome: Percentage of Participants Hospitalized at Least Once Due to a Respiratory Event
Time Frame: Baseline to Day 168
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 61
percentage of participants
  Never hospitalized | 82.0
  Hospitalized at least once | 18.0

7. Secondary Outcome: Number of Days Participants Were Hospitalized Due to a Respiratory Event
Description: The average number of days hospitalized due to a respiratory event, among the 11 participants who were hospitalized for respiratory event, was reported.
Time Frame: Baseline to Day 168
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AZLI
Number analyzed (Participants) | 11
days | 12.6 (8.90)

8. Secondary Outcome: Percentage of Participants With Pulmonary Exacerbations
Description: Pulmonary exacerbations were defined as respiratory hospitalizations or discrete courses of non-study IV/inhaled antipseudomonal antibiotics. Use of oral antibiotics alone for respiratory signs or symptoms was considered to be representative of milder clinical events and, therefore, was not included in the definition of pulmonary exacerbations.
Time Frame: Baseline to Day 168
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 61
percentage of participants
  No pulmonary exacerbation | 62.3
  At least one pulmonary exacerbation | 37.7

9. Secondary Outcome: Time to Pulmonary Exacerbation
Description: The median days to first pulmonary exacerbation was summarized using Kaplan-Meier (KM) summary statistics.
Time Frame: Baseline to Day 168
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI
Number analyzed (Participants) | 61
days | 176.0 [176.0 to NA] — Some participants did not use non-study antipseudomonal antibiotics until the end of the study, so time to non-study antipseudomonal antibiotic use was unknown. Therefore, the upper limit of the 95% CI for median time could not be estimated.

10. Secondary Outcome: Percentage of Participants With Study-drug Induced Bronchospasm
Description: Study-drug induced bronchospasm (airway reactivity) was assessed at the baseline visit as the percent change in FEV1 from the pretreatment measurement to 30 minutes following treatment for subjects ≥ 6 years or as from the Investigator's assessment for subjects < 6 years.
Time Frame: Pretreatment at Baseline to 30 minutes following treatment
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AZLI
Number analyzed (Participants) | 61
percentage of participants | 3.3 (6.06)

11. Secondary Outcome: Adverse Event Rates Adjusted for Study Duration
Description: Adverse events occurring in ≥ 5% of participants adjusted for study duration were summarized. The adjustment was made by using a standardized rate calculated as the sum of study duration across patients divided by 28 for the total number of patient months. Rate calculations presented are the number of adverse events (AEs) per patient month.
Time Frame: Baseline to Day 168
Population: Full Analysis Set
Measure: Number; unit: AEs (per patient month)
Arm/Group | AZLI
Number analyzed (Participants) | 61
AEs (per patient month)
  Cough | 0.163
  Nasal congestion | 0.050
  Rhinorrhoea | 0.041
  Wheezing | 0.033
  Sputum increased | 0.033
  Productive Cough | 0.030
  Lung disorder | 0.025
  Haemoptysis | 0.019
  Rhonchi | 0.019
  Oropharyngeal pain | 0.017
  Rales | 0.017
  Respiratory tract congestion | 0.014
  Abdominal pain | 0.030
  Diarrhoea | 0.019
  Vomiting | 0.019
  Abdominal pain upper | 0.017
  Pyrexia | 0.061
  Fatigue | 0.025
  Rhinitis | 0.030
  Pulmonary function test decreased | 0.014
  Forced expiratory volume decreased | 0.011
  Decreased appetite | 0.017

ADVERSE EVENTS:
Time Frame: Baseline to Day 168
Arm/Group | AZLI
Serious Adverse Events (participants affected / at risk) | 13/61
Other Adverse Events (participants affected / at risk) | 50/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=61)
Appendiceal mucocoele (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gastrointestinal infection (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=61)
Diarrhoea (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 8
Pyrexia (General disorders) | 16
Rhinitis (Infections and infestations) | 10
Pulmonary function test decreased (Investigations) | 5
Forced expiratory volume decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 6
Rales (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years